CLINICAL TRIAL: NCT02788318
Title: Serotoninergic Pathways in Sudden and Unexpted Death in Epilepsy (SUDEP)
Acronym: SUDEP
Status: Terminated | Type: Observational
Why Stopped: difficulty recruiting patients
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: D50830
Record Dates: First submitted 2016-05-27; First posted 2016-06-02 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Sudden Unexpected Death in Epilepsy (SUDEP)
Keywords: Epilepsy; SUDEP; Serotonin
MeSH Terms: conditions — Sudden Unexpected Death in Epilepsy; Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Brain tissue (brainstem, hippocampus and insula) and fibroblasts culture
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- diagnostic of SUDEP: patient with epilepsy in whom anamnestic and post-mortem evidence does not identify a particular cause (diagnosis of SUDEP). Brain samples and skin samples are collected.
  Interventions: Other: Brain samples; Other: Skin samples
- Control 1: Subjects with a known epilepsy, whose death is linked to a specific cause. Brain samples and skin samples are collected.
  Interventions: Other: Brain samples; Other: Skin samples
- Control 2: Subjects without known pathological history, remained victims of unexplained sudden unexpected death (SUDEP) after all investigations and for which a heart rhythm disorder is suspected in first intention. Brain samples and skin samples are collected.
  Interventions: Other: Brain samples; Other: Skin samples

INTERVENTIONS:
Other: Brain samples — Collected in patients died
Other: Skin samples — Collected in patients died

SUMMARY:
The mortality rate is increased in patients with epilepsy, and especially among patients with drug-resistant epilepsy. This increased mortality is mainly related to the risk of SUDEP whose incidence is between 3.5 and 9 per 1,000 for patients with drug-resistant epilepsy. The term SUDEP refers to a sudden death occurring in a patient with epilepsy in whom anamnestic and post-mortem evidence does not identify a particular cause. Experimental and clinical data strongly suggest that most of SUDEP result from a postictal respiratory dysfunction progressing to terminal apnea. Due to the major role of serotonin in regulating breathing rhythms and data in animal models of epilepsy, it is envisaged that an alteration of serotonergic systems of the brainstem and limbic regions may play a central role in the occurrence of SUDEP. The objective of this work is to look for abnormalities of the serotonergic transmission within regulatory regions of respiratory and autonomic functions in brain samples prospectively collected in patients died from SUDEP.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Postmortem time before autopsy <30 hours

Exclusion Criteria:

* Age <18 years
* postmortem time before autopsy > 30 hours
* Any subject whose brain would be of forensic interest
* Any patient who expressed an opposition to organ donation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with epilepsy who died
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Density of Medullary 5-HT Neurons | between 1 to 30 hours following death
  5-HT1A receptor binding density in within the medulla

SECONDARY OUTCOMES:
Other markers of 5HT within the medulla | between 1 to 30 hours following death
  Expression of 5HT-1A and 5HT-2 receptors, expression of 5HT transporter, Tryptophan Hydroxylase 2 (TPH2)
Serotoninergic pathway in the pons, the hippocampus and the insula | between 1 to 30 hours following death
  5-HT1A receptor binding density, Expression of 5HT-1A and 5HT-2 receptors, expression of 5HT transporter, Tryptophan Hydroxylase 2 (TPH2)
Catecholaminergic pathway | between 1 to 30 hours following death
  Number of neurons expressing the tyrosine hydroxylase, expression of alpha and beta adrenergic receptors, expression of dopamine-bêta-hydroxylase

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon - Institut Médico-Légal, Lyon, France